CLINICAL TRIAL: NCT01787903
Title: The Effects of Real-time Continuous Glucose Monitoring on Glycemia and Quality of Life in Patients With Type 1 Diabetes Mellitus and Impaired Hypoglycemia Awareness
Brief Title: The Effects of RT-CGM on Glycemia and QoL in Patients With T1DM and IHA
Acronym: INCONTROL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Erik Serne, MD PhD, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DC2012INCONTROL01
Record Dates: First submitted 2013-02-06; First posted 2013-02-11 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Type 1 Diabetes Mellitus; Hypoglycemia Unawareness
Keywords: Type 1 diabetes mellitus; Hypoglycemia unawareness; Real-time continuous glucose monitoring; Glucose control
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real-time continuous glucose monitor (Active Comparator): 16 weeks use of a real-time continuous glucose monitor
  Interventions: Device: Real-time continuous glucose monitor
- Continuous glucose monitor (Placebo Comparator): 16 weeks use of a (blinded, retrospective) continuous glucose monitor
  Interventions: Device: Real-time continuous glucose monitor

INTERVENTIONS:
Device: Real-time continuous glucose monitor — Active Comparator: MiniMed Paradigm® Veo™-system Placebo Comparator: iPro™2 Continuous Glucose Monitor (masked)
  Other Names: MiniMed Paradigm® Veo™-system; iPro™2 Continuous Glucose Monitor

SUMMARY:
The purpose of this study is to determine what the effects are of real-time continuous glucose monitoring on glycemia and quality of life in patients with type 1 diabetes mellitus and impaired hypoglycemia awareness.

DETAILED DESCRIPTION:
The investigators hypothesize that the use of RT-CGM, relative to a control intervention using masked CGM, will result in improvement of various measures of glycemia and indicators of quality of life, reduce the occurrence of hypoglycemia and hyperglycemia and restore hypoglycemia awareness in T1DM patients with IHA. We will test this hypothesis by addressing the following research questions:

What is the effect of 16 weeks of RT-CGM use, versus 16 weeks of CGM use, in patients with T1DM and IHA on

1. (primary objective:) time spent in euglycemia
2. (secondary objectives:)

   * (diabetes-specific) markers of QoL, covering diabetes-related emotional distress (PAID-5), fear of hypoglycemia (HFS-2), self-efficacy (CIDS), health status (EQ5D) and emotional well-being (WHO-5)
   * other glycemia variables, including HbA1c and time spent in hypo- and - hyperglycemia ranges
   * the incidence and duration of hypoglycemic episodes
   * changes in hypoglycemia awareness score according to Gold et al.,
3. (tertiary objectives:)

   * measures of glucose variability
   * the autonomic nervous system balance
   * the duration of wear of the RT-CGM device
   * patients' therapy adjustments during the interventions
   * hypoglycemia awareness scores according to Clarke et al.
   * satisfaction with use of CGM
   * the number of contact moments not planned according to the study schedule
   * absence of work of patient (and spouse)
   * the global estimated costs of use of health care

ELIGIBILITY:
Inclusion Criteria:

* T1DM, diagnosed according to ADA criteria regardless duration
* Use of multiple daily injections of insulin (with a basal insulin injection and bolus injections) or continuous subcutaneous insulin infusion
* Any HbA1c
* Age between 18 and 70 years old (inclusive)
* IHA according to the questionnaire by Gold et al.
* Performing at least 3 SMBG/day or 21 SMBG/week

Exclusion Criteria:

* Type 2 diabetes mellitus
* History of (recent) major renal, liver, or (ischemic) heart disease (including cardiac conduction disorders)
* Current untreated proliferative diabetic retinopathy
* Current (treatment for) malignancy
* Current use of non-selective beta-blockers
* Current psychiatric disorders, including schizophrenia, bipolar disorder, anorexia nervosa or bulimia nervosa
* Substance abuse or alcohol abuse (men >21 units/week, women >14 units/week)
* Current pregnancy or intention to conceive
* Current use of RT-CGM other than for short term (i.e. diagnostic use or use shorter than 3 consecutive months)
* Hearing or vision impairment hindering perceiving of glucose display and alarms, or otherwise incapable of using a (RT-)CGM, in the opinion of the investigator
* Poor commandment of the Dutch language or any (mental) disorder that precludes full understanding of the purpose and instructions of the study
* Participation in another clinical study
* Known or suspected allergy to trial product or related products

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2013-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Time spent in the euglycemic range | 45 weeks
  The mean difference in time spent in the euglycemic range (interstitial glucose >3.9-<10.0 mmol/L), expressed as hours/day between the two 16-week intervention periods, i.e. RT-CGM versus masked CGM in patients with T1DM and IHA.

SECONDARY OUTCOMES:
Quality of life | 45 weeks
  (diabetes-specific) markers of QoL, covering diabetes-related emotional distress (PAID-5), fear of hypoglycemia (HFS-2), self-efficacy (CIDS), health status (EQ5D) and emotional well-being (WHO-5)
Glycemia variables | 45 weeks
  Other glycemia variables, including HbA1c and time spent in hypo- and hyperglycemia ranges
Hypoglycemic episodes | 45 weeks
  The incidence and duration of hypoglycemic episodes
Changes in hypoglycemia awareness score | 45 weeks
  Changes in hypoglycemia awareness score according to Gold et al.

OTHER OUTCOMES:
Glucose variability | 45 weeks
  RT-CGM derived measures of glucose variability, e.g. SD, MODD, CONGA
ANS balance | 45 weeks
  The autonomic nervous system balance
Sensor wear duration | 45 weeks
  The duration of wear of the RT-CGM device
Therapy adjustments | 45 weeks
  The therapy adjustments made by patients during the interventions
Hypoglycemia awareness score | 45 weeks
  Hypoglycemia awareness scores according to Clarke et al.
RT-CGM satisfaction | 45 weeks
  Satisfaction with use of CGM

CONTACTS AND LOCATIONS:
Overall Officials: Erik H Serné, MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] van Beers CA, DeVries JH, Kleijer SJ, Smits MM, Geelhoed-Duijvestijn PH, Kramer MH, Diamant M, Snoek FJ, Serne EH. Continuous glucose monitoring for patients with type 1 diabetes and impaired awareness of hypoglycaemia (IN CONTROL): a randomised, open-label, crossover trial. Lancet Diabetes Endocrinol. 2016 Nov;4(11):893-902. doi: 10.1016/S2213-8587(16)30193-0. Epub 2016 Sep 15. PMID 27641781
- [Derived] van Beers CA, Kleijer SJ, Serne EH, Geelhoed-Duijvestijn PH, Snoek FJ, Kramer MH, Diamant M. Design and rationale of the IN CONTROL trial: the effects of real-time continuous glucose monitoring on glycemia and quality of life in patients with type 1 diabetes mellitus and impaired awareness of hypoglycemia. BMC Endocr Disord. 2015 Aug 21;15:42. doi: 10.1186/s12902-015-0040-3. PMID 26292721